CLINICAL TRIAL: NCT04069468
Title: A Prospective, Post Approval, Multiple Centre, Open-Label, Non-Interventional, Registry Study to Evaluate Effectiveness of TheraSphere® in Clinical Practice in France
Brief Title: Non-Interventional Registry Study to Evaluate the Effectiveness of TheraSphere® in the Treatment of Hepatocellular Carcinoma (HCC)
Acronym: PROACTIF
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: Biocompatibles UK Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BTG-007996-01
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Prospective Registry; TheraSphere®; France; SIRT; Liver Cancer, Adult; Liver Cell Carcinoma; Hepatoma; Intra arterial treatment; Intra hepatic Cholangiocarcinoma; Colon cancer metastasis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TheraSphere®: Patients with HCC, iCC and mCRC will be treated. TheraSphere is administered in the liver through the hepatic artery. Treatment will be performed according to the Instructions for Use (IFU). Activity of administered TheraSphere is tailored in order to deliver an absorbed dose of 80 to150 gray (Gy) to the liver. Lung dose (D) will be calculated from the following formula: D=A*(1-S)*50/1. D=Planned dose absorbed by treated volume(Gy), A=Activity injected with microspheres (gigabequerel [GBq]), S=Percentage of pulmonary shunt, "1" assuming that the lung mass=1 kilograms [kg]). Number of treatments is up to Investigator's discretion while taking into account the cumulative dose to the liver and lung.
  Interventions: Device: TheraSphere

INTERVENTIONS:
Device: TheraSphere — Participants will receive treatment with TheraSphere in accordance with Instructions for Use
  Other Names: Yttrium-90 Glass Microspheres

SUMMARY:
The purpose of this registry study is to gather effectiveness, QoL, safety and procedural information on TheraSphere® for the treatment of participants with Hepatocellular Carcinoma (HCC), Intrahepatic Cholangiocarcinoma (iCC) and liver metastases for colon cancer (mCRC) in real world clinical practice settings in France.

DETAILED DESCRIPTION:
TheraSphere is a radioembolic therapeutic device used in the treatment of liver cancers. The goal of the registry study is to collect prospectively: participant description, treatment goal, treatment description, treatment results, safety, quality of life and survival data to ultimately demonstrate that TheraSphere treatment meets the claims that led to the reimbursement in France. The registry study is also an opportunity to improve the proper use of the device by team training especially for the personalized dosimetry treatment approach.

Clinical data will be collected and held in a secured, validated system and can be downloaded by Biocomplatibles UK Ltd Data Management on an ongoing basis. Data verification will be performed by Biocompatibles UK Ltd Data Management and data validation checks will be created by the validated data system (with the Biocompatibles UK Ltd team performing User Acceptance Testing on them before they go live). Adverse Events and concomitant diseases will be coded according to the version of Medical Dictionary for Regulatory Activities (MedDRA) agreed with Biocompatibles UK Ltd. Concomitant medications will be coded using the version of the World Health Organisation (WHO) Drug dictionary agreed with the validated data system.

Appropriate study plans implemented to manage all aspects of the trial to ensure quality and integrity of the data collection.

ELIGIBILITY:
Inclusion:

* Participant has received a reimbursed dose of TheraSphere®
* Participant does not oppose to the collection of his/her medical personal data

Exclusion:

* Participant has opposed to data collection
* Participant has not received a reimbursed dose of TheraSphere® (free of charge dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants for whom treatment with TheraSphere® has been prescribed and reimbursed in France will be eligible for this study. It is estimated that data from >500 participants will be entered into this registry from approximately 30 sites in France.
Sampling Method: Non-Probability Sample
Enrollment: 1247 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Treatment (Day 1) up to participant's death, opposition to data collection, or study termination (up to Year 6)
  OS will be calculated as the interval between treatment administration and the date of death for any cause, opposition to data collection, or study termination, whichever occurs first.
QoL Measurements Using FACT-HEP Questionnaire Before and After Treatment | Treatment (Day 1), every 2 to 4 months Post Treatment (maximum treatment time = up to Day 28), and SOC visits after Month 12 until up to participant's death, opposition to data collection, study withdraw for any cause, or study termination (up to Year 6)
  Quality of Life (QoL) will be assessed by the Functional Assessment of Cancer Therapy (FACT-HEP) questionnaire prior to treatment on Day 1, every 2 to 4 months post treatment (follow up visits), and every standard of care (SOC) visit after Month 12 until the participant's death, opposition to data collection, study withdraw for any cause, or study termination. The FACT-Hep Questionnaire uses participant-reported outcome (PRO) scores. QoL scores of each domain at each time-point and their differences from baseline will be summarised. A deterioration in QoL is defined as a 7-point decline in the total score or death, whichever comes first. The time to deterioration in QoL will be calculated as the interval between first date of TheraSphere® treatment and deterioration in QoL. The higher the score, the better the QoL, with a range 0-180.

SECONDARY OUTCOMES:
Number of Grade 3 or Higher Adverse Events (AEs) Related to Study treatment or Procedure | Treatment (Day 1) up to 90 Days Post Treatment or the first post treatment follow-up visit after TheraSphere administration, if after 90 days (maximum treatment time = up to Day 28)
  An AE is any untoward medical occurrence or undesirable event experienced in a participant that begins or worsens following TheraSphere® administration. AEs will be classified using National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v 5.0.
Number of Participants Re-Hospitalised Following Treatment | Treatment (Day 1) up to Month 1 Post Treatment (maximum treatment time = up to Day 28)
  The number of participants re-hospitalised for any event related to TheraSphere® treatment during the study will be reported.
Duration of Re-Hospitalisations Following Treatment | Treatment (Day 1) up to Month 1 Post Treatment (maximum treatment time = up to Day 28)
  The duration of re-hospitalisations for any event related to TheraSphere® treatment during the study will be reported.
Number of Participants Achieving Treatment Expectation | Baseline up to Month 12 Post Treatment
  At Baseline and follow-up post treatment, participants' treatment expectation will be measured by a qualitative assessment according to Investigator's opinion, whether the goal is met or not. Before treatment the treatment goal will be documented. The number of participants achieving the treatment goal will be reported.
Number of Participants with Tumour Response | Treatment (Day 1) up to Month 12 Post Treatment (maximum treatment time = up to Day 28)
  Tumour Response will be based on the radiological tumour assessment and will be categorized as Complete Response (CR), Partial Response (PR), Stable Disease (SD) or Progressive Disease (PD). Tumour response will be assessed using Modified Response Evaluation Criteria in Solid Tumours (mRECIST) criteria or RECIST criteria
Number of Participants with an Alpha-Fetoprotein (AFP), CA 19-9, CEA tumour Response | Treatment (Day 1) and Month 12 Post Treatment (maximum treatment time = up to Day 28)
  A Tumour response defined as a ≥50% decrease in: AFP levels for participants with a Baseline AFP level ≥200 nanograms/milliliter (ng/mL), CA 19-9 levels for participants with a baseline CA 19-9 level ≥ 2 x Upper Limit of Normal (ULN), CEA levels for participants with a baseline CEA level ≥ 2 x ULN.
Number of Participants Receiving a Post TheraSphere Anti-Cancer Treatment | Treatment (Day 1) up to participant's death, opposition to data collection, study withdraw for any cause, or study termination (up to Year 6)
  The number of participants for which additional TheraSphere treatment or surgical procedure is required will be reported.
Number of Participants Reporting Best Supportive Care Treatment | Treatment (Day 1) up to participant's death, opposition to data collection, study withdraw for any cause, or study termination (up to Year 6)
  The number of participants for which additional anti-cancer treatment including additional TheraSphere treatment or surgical procedure will be reported.
Number of Participants per Type of Vascular Access Used to Administer TheraSphere | Treatment (Day1) upto Month 12
  The number of participants recorded for each type of vascular access (that is, Femoral/Radial-Humeral) will be reported.
Number of Participants with similar Tumour(s) Location at Baseline and the location of lesions targeted by 99mTc-MAA SPECT Imaging | Baseline and Post 99mTc-MAA Imaging (up to Day 28)
  The Baseline computed tomography (CT)/magnetic resonance imaging (MRI) will be compared against 99mTc-MAA imaging (Single Proton Emission Computed Tomography [SPECT] or SPECT/CT) to evaluate the agreement in the lesion locations identified with 2 imaging methods. The 3 categories to report agreement between Baseline CT/MRI and 99mTc-MAA are: Optimal (images match), Sub optimal (less than 50% matching), and Non optimal (images do not match at all).
Description of post treatment tumour targeting by determination of the number of patients with similar tumour(s) location at baseline and location of lesions targeted by Y-90 Positron Emission Tomography (PET)/CT or Y-90 PET/MRI or Y-90 SPECT/CT. | Baseline and Post TheraSphere Administration Imaging (up to Day 28)
  The Baseline CT/MRI will be compared against the Post TheraSphere administration imaging (Y90-SPECT-CT, or Y90-PET-CT, or Y90-PET-MRI) to measure agreement in the lesion locations identified with the 2 imaging methods. The 3 categories to evaluate the agreement between Baseline CT/MRI and 99mTc-MAA are: Optimal (images match), Sub optimal (less than 50% matching), and Non optimal (images do not match at all).
Description of pre and post treatment tumour targeting by determination of the number of patients with similar tumour(s) location based on 99mTc-MAA (SPECT or SPECT/CT and location of tumour targeted by Y-90 using post-treatment(PET/CT or PET/MRI or SPEC | Pre-Treatment Administration (Baseline) and Post-Treatment Administration (up to Day 28)
  99mTc-MAA SPECT-CT will be compared against the Post TheraSphere administration (Y90-SPECT-CT, or Y90-PET-CT, or Y90-PET-MRI) to measure agreement in the lesion locations identified with the 2 imaging methods. The 3 categories to report agreement between Baseline 99mTc-MAA SPECT-CT and TheraSphere (Y90-SPECT-CT, or Y90-PET-CT, or Y90-PET-MRI) are: Optimal (images match), Sub optimal (less than 50% matching), and Non optimal (images do not match at all).
Description of Portal Vein Thrombosis (PVT) targeting by determination of the number of patients with PVT at baseline that have the PVT targeted by 99mTc-MAA (SPECT or SPECT/CT), Y-90 (PET/CT or PET/MRI or SPECT/CT). | Pre-Treatment Administration (Baseline) and Post-Treatment Administration (up to Day 28)
  Types of PVT will be classified according to the following scale: Vp0 Absent; Vp1 Presence or tumour thrombus distal to, but not in, the second-order branches of the portal vein; Vp2 Presence of tumour thrombus in first -order branches of the portal vein; Vp3 Presence of tumour thrombus in first-order branches of the portal vein; and Vp4 Presence of tumour thrombus in the main trunk of portal vein or a portal vein contralateral to the primary involved lobe (or both). In case of PVT (Vp1 to Vp4), the intensity of 99mTc-MAA and TheraSphere uptake on PVT (that is, greater activity than surrounding treated liver parenchyma) evaluated on 99mTc-MAA SPECT-CT, Y90-SPECT-CT, or Y90-PET-CT or Y90-PET-MRI imagings will be graded qualitatively as strong, weak or no uptake on PVT.
Determination of a correlation between tumour and normal tissue liver absorbed doses, determined with 99mTc-MAA (SPECT or SPECT/CT), with qualitative tumour response (CR or PR), OS and safety, respectively as Assessed by Cox Regression Analyses | Baseline and Post 99mTc-MAA Imaging (up to Day 28)
  A Cox regression analysis of OS will be performed to assess the impact of the tumour and normal liver tissue absorbed doses. This will be done separately for absorbed doses calculated before treatment administration with 99mTc-MAA (SPECT or SPECT/ CT) and estimated with post-treatment TheraSphere Y90-PET-CT or Y90-PET-MRI.
Determination of a correlation between tumour and normal tissue liver absorbed doses, determined with Y-90 (PET/CT or PET/MRI), with qualitative tumour response (CR or PR), OS and safety, respectively. | Baseline and Post 99mTc-MAA Imaging (up to Day 28)
  A logistic regression analysis of qualitative tumour/index lesion response (CR or PR) will be performed to assess the impact of the tumour/index lesion AD (i.e. the response variable is whether there was a response and the explanatory variable is the AD). This will be done separately for ADs from pre-procedural 99mTc-MAA (SPECT or SPECT/CT) and for post-procedural Y-90 PET/CT or PET/MRI. A Cox regression analyses of OS will be performed to assess the impact of the tumour ADs (i.e., the AD will be the explanatory variable). This will be done separately for AD by 99mTc-MAA (SPECT or SPECT/CT) and by post-treatment Y-90 PET/CT and/or PET/MRI. Logistic regression analyses of the occurrence of SAEs will be performed to assess the impact of the non-tumoural liver absorbed doses. This will be done separately for absorbed doses calculated before treatment administration with 99mTc-MAA (SPECT or SPECT/ CT) and estimated with post-treatment TheraSphere® Y90-PET-CT or Y90-PET-MRI
Determination of a correlation between tumour and normal tissue liver absorbed doses determined with 99mTc-MAA (SPECT or SPECT/CT) and with Y-90 (PET/CT or PET/MRI) | Baseline and Post 99mTc-MAA Imaging (up to Day 28)
  The relationship between absorbed doses derived from pre-procedural 99mTc-MAA (SPECT or SPECT/CT) imaging and post-treatment Y90 PET/CT or PET/MRI imaging will be assessed separately for normal tissue liver absorbed doses and tumour absorbed doses using Bland-Altman analysis.
Determination of a correlation between Dose volume histogram (DVH) for total perfused tumour, Index lesion and whole normal liver tissue, using 99mTc-MAA (SPECT or SPECT/CT) and Y-90 (PET/CT or PET/MRI). | Baseline and Post 99mTc-MAA Imaging (up to Day 28)
  The DVH using 99Tc-MAA and TheraSphere (Y90-SPECT-CT, Y90-PET-CT, or Y90-PET-MRI) will be reported for total perfused tumours, index lesions, and whole normal liver tissues. The observed counts will be presented. A linear regression of AD from pre-procedural 99mTc-MAA (SPECT or SPECT/CT) imaging and post-procedural Y-90 PET/CT or PET/MRI imaging will be performed and Pearson's correlation coefficient will be calculated.

CONTACTS AND LOCATIONS:
Locations (37):
- France (37):
  - CHU Amiens, Amiens
  - CHU, Angers, Angers
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Hôpital Haut Leveque, Bordeaux
  - Centre Hospitalier Régional et Universitaire de Brest, Brest
  - Hôpital Henri Mondor, Créteil
  - Centre George-Francois Leclerc, Dijon
  - CHU Dijon Bourgogne, Dijon
  - CHU Michallon, Grenoble
  - Bicêtre Hôpital, Le Kremlin-Bicêtre
  - CHU Lille, Lille
  - Centre Leon Berard, Lyon
  - Hopital de la Croix-Rousse, Lyon
  - Hopital Edouard Herriot, Lyon
  - CHU de la Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - CHU Saint Eloi, Montpellier
  - CHU Brabois Adultes, Nancy
  - CHU Site Hotel Dieu, Nantes
  - CHU de l'Archet, Nice
  - CHU de Nîmes, Hôpital Carremeau, Nîmes
  - Hopital Beaujon, Paris
  - Hôpital Cochin, APHP, Paris
  - Hôpital Saint-Louis, Paris
  - Centre Hospitalier de Perpignan, Perpignan
  - Hopital Lyon Sud, Pierre-Bénite
  - CHU La Milétrie, Poitiers
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU Rouen, Rouen
  - Centre Hospitalier Universitaire de St Etienne, Saint-Priest-en-Jarez
  - CHU deHautepierre, Strasbourg
  - Nouvel Hopital Civil, Strasbourg
  - CHU Rangueil, Toulouse
  - Hopital Paul Brousse, Villejuif
  - Intstitut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Garin E, Pinaquy JB, Bailly C, Sengel C, Mariano-Goulart D, Edeline J, Blanc JF, Bouvier A, Tordo J, Rode A, Becker S, Sefrioui D, de Baere T, Somma C, Mastier C, Goupil J, Chevallier P, Regnault H, Vibert E, Manfredi S, Vicaut E, Patel B, Boucher E, Guiu B; PROACTIF registry group. Evaluating the Effectiveness of Yttrium-90 Glass Microspheres in the Treatment of Hepatocellular Carcinoma, Intrahepatic Cholangiocarcinoma, and Metastatic Colorectal Cancer in Practice: Protocol for the Prospective PROACTIF Phase IV Registry Study in France. Cardiovasc Intervent Radiol. 2022 Jan;45(1):1-11. doi: 10.1007/s00270-021-03002-0. Epub 2021 Nov 18. PMID 34796373